CLINICAL TRIAL: NCT05276232
Title: Detection of Cannabis Impairment With ISBRG's SpotLight-THC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ISBRG Corp (Other)
Collaborators: National Advanced Driving Simulator (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202108451
Record Dates: First submitted 2022-02-11; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Cannabis
Keywords: Driving under the influence; Cannabis impairment; SpotLight-THC; Non-invasive detection; THC; ISBRG
MeSH Terms: conditions — Marijuana Abuse; Driving Under the Influence | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baseline followed by 5-10% THC Validation (Experimental)
  Interventions: Drug: Cannabis(THC) inhaled
- Baseline followed by 5-10% THC Verification (Experimental)
  Interventions: Drug: Cannabis(THC) inhaled

INTERVENTIONS:
Drug: Cannabis(THC) inhaled — Cannabis vapor is produced from 500mg, approximately 5-10% High dose bulk cannabis plant material, 30-37.5 mg THC

SUMMARY:
Subjects will participate in a 2-visit study protocol in which they will be administered cannabis of pre-determined concentrations and asked to complete a simulated drive in a driving simulator. Subjects will be scanned on two SpotLight-THC (Alpha and Beta iterations) devices and peripheral venous whole blood will be collected from subjects for analysis on up to four occasions on each visit.

The purpose of the investigation will be to determine whether the SpotLight-THC device is a reliable measure of THC impairment at the roadside, with an objective to identify a unique blood analyte architecture for THC impairment using near infrared light and machine learning.

DETAILED DESCRIPTION:
At the University of Iowa, subjects who currently use cannabis recreationally will be recruited. They will then undergo a screening visit in which consent is obtained, questionnaires are given, a physical exam is conducted and subjects will use the driving simulator to assess propensity to sickness and to familiarize them with the simulation. They will then be scheduled for their next visit. At the second visit, subjects will be administered 5-10% THC. A series of baseline tests, including a test requiring a blood sample will be administered upon arrival. After drug administration, subjects will be asked to complete a set of verbal recall questions followed by three simulated driving trials, completing 7 non-invasive SpotLight-19 scans (20 seconds x 2) and 3 blood samples throughout the visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged at least 18 years old
* Must self-report use of cannabis at least once a month
* Has held a valid driver's license at least 12 months
* Must be willing to abstain from using cannabis and alcohol for 24 hours prior to each session
* Must be willing to abstain from all other drugs not medically required for duration of the study (beginning 24 hours prior to the screening visit)
* Must be able to drive without special or non-standard equipment
* Must be able to meet study time commitment
* Provides written and informed consent

Exclusion Criteria:

* Diagnosis of severe medical or psychiatric condition (as judged by study physician)
* Evidence of substance use disorder as reflected by total scores on DUDIT and AUDIT
* Regular user of medication that may affect cognitive functioning and/or driver performance (e.g., antidepressants, benzodiazepines, stimulants, opioids) as judged by study physician
* Family history of schizophrenia or other psychotic disorder (or taking medications for such)
* Pregnant or test positive for pregnancy, looking to become pregnant, or breastfeeding
* Respiratory or pulmonary disorder that would negatively affect ability to inhale and hold the cannabis dose
* Recent (past 6 months) head injury or stroke, or current symptoms from prior head injury or stroke
* History of heart disease, angina, heart attack, heart surgery, or myocardial infarction (or taking medications for such)
* Untreated/Untreatable vision or auditory issues (because testing currently requires both senses)
* History of suicidal behaviors in past two years
* Excessive tobacco use (more than 10 cigarettes a day or 3 or more cigars or pipes per day)
* Excessive caffeine use (6 or more servings per day)
* Excessive alcohol (14 or more drinks per week)
* Regular use of pain medications other than OTC
* Use of prescription drugs not prescribed to them or illicit drugs other than cannabis
* History of substance abuse or substance addiction
* Expressed interest in or participation in drug abuse treatment in past 60 days
* Currently diagnosed cannabis use disorder
* History of negative reaction to cannabis
* Extreme scarring on fingertips that prevents use of the device
* Participation in night shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in Acute Subjective Response to Cannabis Score | At baseline, 20, 30, 60, 90, 120 and 180 minutes
  The total score of the true responses (true/false scale, minimum score is 0 with a maximum score of 12). A higher score indicates greater drug effect. Used to determine subjective level of drug effect.

SECONDARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) - Undistracted | Over a 20 minute drive conducted at 30, 90 and 180 minutes post dose
  The ability to keep the vehicle straight in the lane and the corresponding data is presented from a rural drive without any secondary tasks relative to the 20 minute baseline drive pre dose.
Standard Deviation of Lateral Position (SDLP) - Distracted | Over a 20 minute drive conducted at 30, 90 and 180 minutes post dose
  The ability to keep the vehicle straight in the lane and the corresponding data is presented from a rural drive while engaged in a secondary task relative to the 20 minute baseline drive while engaged in the same task pre dose.
Blood Delta-9-THC | At baseline, 20, 90, and 180 minutes
  THC concentration levels of Delta-9-THC in whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Brown, Ph.D., Principal Investigator — National Advanced Driving Simulator
Locations (1):
- National Advanced Driving Simulator, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No